CLINICAL TRIAL: NCT00464932
Title: Vasoactive Intestinal Peptide in COPD
Acronym: VIPCOPD
Status: Completed | Type: Observational
Sponsor: Medical University of Vienna (Other)
Other Study IDs: EK 168/2003
Record Dates: First submitted 2007-04-23; First posted 2007-04-24 (Estimated); Last update posted 2007-04-24 (Estimated); Status verified 2007-04

CONDITIONS: COPD; Pulmonary Hypertension
Keywords: COPD; Vasoactive Intestinal Peptide; Lung Function
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Hypertension, Pulmonary | interventions — Vasoactive Intestinal Peptide

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Vasoactive Intestinal Peptide (VIP)

SUMMARY:
This study, a new immunomodulatory therapy of COPD with vasoactive intestinal peptide (VIP) was evaluated. Based on preliminary unpublished clinical and experimental results, the course of disease under VIP treatment and the molecular mechanisms involved were assessed.

34 patients with severe COPD were treated either with VIP inhalation in addition to conventional therapy or inhalation of placebo plus conventional therapy for a period of 3 months. The trial was conducted as a double blind, comparative study with two parallel groups.

DETAILED DESCRIPTION:
Chronic obstructive bronchitis is a chronic inflammatory disease of the airways, which affects as many as 8% of individuals in industrialized nations. There is an increase in the number of woman and men suffering from COPD. Pulmonary hypertension and cor pulmonale are common sequelae of chronic airflow obstruction, but the precise mechanisms of increased vascular resistance are unclear. Potential causes of pulmo-nary hypertension in COPD include emphysematous destruction of the capillary bed, remodeling of pulmonary vessels and hypoxic pulmonary vasoconstriction. This proposal, a new immunomodulatory therapy of COPD with vasoactive intestinal peptide (VIP) was evaluated. Based on preliminary unpublished clinical and experimental results, the course of disease under VIP treatment and the molecular mechanisms involved were assessed.

34 patients with severe COPD were treated either with VIP inhalation in addition to conventional therapy or inhalation of placebo plus conventional therapy for a period of 3 months. The trial was conducted as a double blind, comparative study with two parallel groups.

In the absence of acute infection or acute worsening of the disease due to other conditions, 2 transbronchial biopsies were collected before treatment, and after 3 months of treat¬ment for assessment of the regulation of a) the immune response, b) the extracellular matrix and c) the epithelial growth. This assessment will be performed in fully equipped and experienced laboratories at the University of Vienna.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed moderate to severe COPD with or without pulmonary hypertension
* Male and female patients.
* Aged 18 - 75 years.
* Written consent.
* Adequate contraception in female patients of childbearing age.
* Negative pregnancy test (four-weekly test repetition).

Exclusion Criteria:

* Lack of consent
* Pregnancy (four-weekly tests)
* Lactation
* Presumed non-cooperativeness
* Patients outside the stipulated age range
* Myocardial infarction within the last 12 months
* Stroke within the last 12 months
* Malignant diseases in anamnesis
* Legal incapacity
* Parallel participation in a clinical trial
* Parallel participation in a clinical trial within the last 4 weeks

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34
Dates: Start 2003-06; Study Completion 2006-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lutz-Henning Block, MD, Principal Investigator — Medical University of Vienna, Department of Pulmology